CLINICAL TRIAL: NCT05982340
Title: Endogenous Lithium Clearance in Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 03055 PVO
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury Due to Sepsis; Proximal Tubule Function; Lithium Clearance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: ICU patients with AKI
  Interventions: Diagnostic Test: Lithium clearance
- Group 2: ICU patients with normal renal function
  Interventions: Diagnostic Test: Lithium clearance

INTERVENTIONS:
Diagnostic Test: Lithium clearance — Blood and urine samples

SUMMARY:
Critically ill patients are at high risk of developing acute kidney injury (AKI). Lithium is freely filtrated at the glomerulus and almost completely reabsorbed in the proximal tubule, which provides a quantitative estimation of proximal tubule reabsorption. The investigators hypothesized that endogenous lithium reabsorption is impaired in the early stages of critical illness.

Investigators would like to study 10 ICU patients with AKI diagnosed, 10 patients without AKI, and 10 healthy controls.

DETAILED DESCRIPTION:
Blood and urine samples will be obtained at 08:00, 14:00 and 20:00 during one day. Renal clearance of creatinine (CCr) and lithium will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients diagnosed with AKI, without AKI and healthy controls

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Renal lithium clearance | 2 days
  Clearance of lithium from the body

CONTACTS AND LOCATIONS:
Overall Officials: Lars MG Ytrebø, MD PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No